CLINICAL TRIAL: NCT03745144
Title: A Randomized, Double-blind, 2-Period, 2-Sequence Crossover Phase I Study With a 1 Month run-in Period to Examine the Effect of Cladribine Tablets on the PK of a Monophasic Oral Contraceptive Containing Ethinyl Estradiol and Levonorgestrel (Microgynon®) in Pre-Menopausal Women With RMS
Brief Title: Effects of Cladribine Tablets on the PK of Microgynon®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: MS700568_0031; 2018-001015-70 (EudraCT Number); NCT04086225 (obsolete NCT alias)
Record Dates: First submitted 2018-11-14; First posted 2018-11-19 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-08

CONDITIONS: Relapsing Multiple Sclerosis (RMS)
Keywords: Multiple Sclerosis; Cladribine; Microgynon®
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cladribine; ethinyl estradiol, levonorgestrel drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sequence 1: First Cladribine, Then Placebo (Experimental): Period 1: Participants received a single once daily dose of Microgynon® tablet from Day 1-8 followed by 5-day once-daily Cladribine 10 to 20 milligram(mg) depending on body weight along with Microgynon® tablet once daily from Day 9-28.
  Period 2: Participants received a single once daily dose of Microgynon® tablet from Day 1-8 followed by 5-day once-daily Cladribine matched Placebo along with Microgynon® from Day 9-14. From Day 15-28 participants received once daily Microgynon® along with 5-day once-daily Cladribine 10 to 20 mg depending on body weight.
  Interventions: Drug: Cladribine; Drug: Placebo; Drug: Microgynon®
- Sequence 2: First Placebo, Then Cladribine (Experimental): Participants 5-day once daily Period 1: Participants received a single once daily dose of Microgynon® tablet from Day 1-8 followed by 5-day once-daily Cladribine matched Placebo along with Microgynon® tablet once daily from Day 9-28.
  Period 2: Participants received a single once daily dose of Microgynon® tablet from Day 1-8 followed by 5-day once-daily Cladribine 10 to 20 mg depending on body weight along with Microgynon® tablet once daily from Day 9-28.
  Interventions: Drug: Cladribine; Drug: Placebo; Drug: Microgynon®
- Microgynon® (Experimental): Participants received Microgynon® for 21 days, starting on the first day of the menstrual cycle.
  Interventions: Drug: Microgynon®

INTERVENTIONS:
Drug: Cladribine — Participants received cladribine once-daily for 5 consecutive days in treatment period 1 and 2.
  Arms: Sequence 1: First Cladribine, Then Placebo; Sequence 2: First Placebo, Then Cladribine
Drug: Placebo — Participants received placebo matched to cladribine once-daily for 5 consecutive days in treatment period 1 and 2.
  Arms: Sequence 1: First Cladribine, Then Placebo; Sequence 2: First Placebo, Then Cladribine
Drug: Microgynon® — Participants received Microgynon® tablet once daily for 21 days in treatment period 1 and 2. Participants received Microgynon® for 21 days, starting on the first day of the menstrual cycle in Run-in period.

SUMMARY:
The purpose of this study was to investigate the potential effects of cladribine on the pharmacokinetics (PK) of monophasic oral contraceptive microgynon® by assessment of its constituents, ethinyl estradiol (EE) and levonorgestrel (LNG).

ELIGIBILITY:
Inclusion Criteria:

* Are pre-menopausal women with or without child-bearing potential with a negative serum pregnancy test, and women with child-bearing potential receiving adequate birth control
* Participants with diagnosis of clinically stable and definite relapsing multiple sclerosis (RMS)
* Adequate hematological, hepatic and renal function as defined in the protocol
* Are able and willing to accept dietary restrictions and restrictions regarding the use of concomitant medications (including over-the-counter products, herbal medicines and dietary supplements) over the course of the study
* Had a body weight and body mass index (BMI) within the range at screening
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* History of clinically relevant allergy or known hypersensitivity to the active substance or to any of the excipients of cladribine tablets or hypersensitivity to drugs with a similar chemical structure to cladribine - History of clinically relevant allergy or known hypersensitivity to 1 of the active substances levonorgestrel (LNG) or ethinylestradiol (EE) or to any excipients of Microgynon® tablets
* Positive results from serology examination for Hepatitis B surface antigen (HbsAg) not due to vaccination, hepatitis B core antibody (HbcAb), Hepatitis C virus antibody (anti- HCV) or Human Immunodeficiency antibody (anti-HIV)
* Presence or risk of venous thromboembolism (VTE) arterial thromboembolism (ATE)
* Diabetes mellitus (Type 1 or Type 2) with vascular manifestations
* Signs or symptoms of neurological disease other than multiple sclerosis (MS) that could explain the symptoms of the participant
* Presence of gastrointestinal (GI) disease or history of gastrointestinal -tract surgery
* Exposure to another investigational drug within the last 2 months or within last 6 month if agent is known to be immunosuppressive
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (7):
- Germany (2):
  - St. Josef und St. Elisabeth Hospital gGmbH, Bochum
  - Nuvisan GmbH, Neu-Ulm
- Poland (5):
  - M.A. - LEK A.M.Maciejowscy SC., Katowice
  - BioResearch Group Sp. z o. o, Nadarzyn
  - IKARDIA Hospital Cardiology, Nałęczów
  - BioVirtus Research Site Sp, Otwock
  - MTZ Clinical Research Sp. z o.o., Warsaw

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS700568_0031
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 37 participants were screened, out of which 28 participants enrolled in the study.
Groups:
- Sequence 2: First Placebo, Then Cladribine: Period 1: Participants received a single once daily dose of Microgynon® tablet from Day 1-8 followed by 5-day once-daily Cladribine matched Placebo along with Microgynon® tablet once daily from Day 9-28.
  Period 2: Participants received a single once daily dose of Microgynon® tablet from Day 1-8 followed by 5-day once-daily Cladribine 10 to 20 mg depending on body weight along with Microgynon® tablet once daily from Day 9-28.
Period: Run-in-Period (Day 0 to Day 28)
Arm/Group | Microgynon® | Sequence 1: First Cladribine, Then Placebo | Sequence 2: First Placebo, Then Cladribine
Started | 28 | 0 | 0
Safety Analysis Set (Safety Analysis Set included all participant who were administered any dose of the trial medication.) | 28 | 0 | 0
Pharmacokinetic Analysis Set (Pharmacokinetic Analysis Set included all participants in the Safety Set without clinically important protocol deviations/violations and absence of factors/events likely to affect Pharmacokinetics (PK).) | 21 | 0 | 0
Completed | 24 | 0 | 0
Not Completed | 4 | 0 | 0
Not completed — Other | 4 | 0 | 0
Period: Period 1
Arm/Group | Microgynon® | Sequence 1: First Cladribine, Then Placebo | Sequence 2: First Placebo, Then Cladribine
Started | 0 | 13 | 11
Completed | 0 | 13 | 10
Not Completed | 0 | 0 | 1
Not completed — Other | 0 | 0 | 1
Period: Period 2
Arm/Group | Microgynon® | Sequence 1: First Cladribine, Then Placebo | Sequence 2: First Placebo, Then Cladribine
Started | 0 | 13 | 10
Completed | 0 | 13 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who were administered any dose of the trial medication.
Groups:
- All Participants: All participants who received Microgynon® for 21 days and received cladribine treatment of 10 to 20 mg depending on body weight or matching placebo treatment in either of Treatment groups.
Arm/Group | All Participants
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Zero to Tau at Steady State (AUCt,ss) of Ethinyl Estradiol and Levonorgestrel
Description: Area under the plasma concentration-time curve from zero to tau at steady state (AUCt,ss) of ethinyl estradiol and levonorgestrel were reported. Calculated using descriptive statistics.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post-dose on Day 14
Population: Pharmacokinetic Analysis Set included all participants in the Safety Set without clinically important protocol deviations/violations and absence of factors/events likely to affect Pharmacokinetics (PK).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*picograms per millilitre(h*pg/ml)
Groups:
- Microgynon + Cladribine: Participants received once-daily Cladribine at a dose of 10 milligrams (mg) or 20 mg from Day 9 to Day 13 in period 1 and from Day 15 to Day 19 in Period 2 along with Microgynon® tablet (ethinyl estradiol 30 micrograms [mcg], levonorgestrel 150 mcg) once daily from Day 1 to Day 21 in either treatment period 1 or period 2.
- Microgynon + Placebo: Participants received 5-day once daily cladribine matched placebo from Day 15 to Day 19 in Period 1 and from Day 15 to Day 19 in Period 2 along with Microgynon® tablet (ethinyl estradiol 30 mcg, levonorgestrel 150 mcg) once daily from Day 1 to Day 21 in either treatment period 1 or period 2.
Arm/Group | Microgynon + Cladribine | Microgynon + Placebo
Number analyzed (Participants) | 21 | 21
hour*picograms per millilitre(h*pg/ml)
  Ethinyl Estradiol | 789 (56.9) | 817 (52.6)
  Levonorgestrel | 91400 (45.2) | 92000 (46.8)

2. Primary Outcome: Maximum Observed Plasma Concentration in Steady State (Cmax,ss) of Ethinyl Estradiol And Levonorgestrel
Description: Maximum observed plasma concentration in steady state (Cmax,ss) of ethinyl estradiol and levonorgestrel were reported. Calculated using descriptive statistics.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post-dose on Day 14
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/ml
Arm/Group | Microgynon + Cladribine | Microgynon + Placebo
Number analyzed (Participants) | 21 | 21
pg/ml
  Ethinyl Estradiol | 88.3 (46.5) | 88.1 (45.7)
  Levonorgestrel | 7950 (33.9) | 8150 (34.6)

3. Primary Outcome: Minimum Observed Plasma Concentration in Steady State (Cmin,ss) of Ethinyl Estradiol and Levonorgestrel
Description: Minimum observed plasma concentration in steady state (Cmin,ss) of ethinyl estradiol and levonorgestrel were reported. Calculated from descriptive statistics.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post-dose on Day 14
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/ml
Arm/Group | Microgynon + Cladribine | Microgynon + Placebo
Number analyzed (Participants) | 21 | 21
pg/ml
  Ethinyl Estradiol | 14.8 (66.3) | 14.7 (65.6)
  Levonorgestrel | 2520 (49.5) | 2430 (56.3)

4. Primary Outcome: Plasma Concentration at End of Dosing Interval at Steady State (Ctrough) of Ethinyl Estradiol and Levonorgestrel
Description: Plasma concentration at end of dosing interval at steady state (Ctrough) of ethinyl estradiol and levonorgestrel were reported. Calculated from descriptive statistics.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post-dose on Day 14
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/ml
Arm/Group | Microgynon + Cladribine | Microgynon + Placebo
Number analyzed (Participants) | 21 | 21
pg/ml
  Ethinyl Estradiol | 15.5 (66.8) | 15.4 (66.9)
  Levonorgestrel | 2580 (48.5) | 2580 (56.0)

5. Primary Outcome: Time to Reach the Maximum Observed Plasma Concentration At Steady State (Tmax,ss) of Ethinyl Estradiol and Levonorgestrel
Description: Time to reach the maximum observed plasma concentration at steady state (Tmax,ss) of Ethinyl Estradiol and Levonorgestrel were reported. Calculated using descriptive statistics.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post-dose on Day 14
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Microgynon + Cladribine | Microgynon + Placebo
Number analyzed (Participants) | 21 | 21
hours
  Ethinyl Estradiol | 1.00 [0 to 2.00] | 1.00 [0.417 to 2.00]
  Levonorgestrel | 1.00 [0.417 to 2.00] | 1.00 [0.417 to 2.00]

6. Primary Outcome: Average Plasma Concentration at Steady State (Cav,ss) of Ethinyl Estradiol and Levonorgestrel
Description: Average plasma concentration at steady state (Cav,ss) ) of Ethinyl Estradiol and Levonorgestrel were reported. Cav,ss =AUCt,ss/ tau, where, AUCt,ss was defined as the area under the plasma concentration-time curve in steady state during a complete dosing interval (tau) and Tau is the Complete dosing interval. Calculated using descriptive statistics.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post-dose on Day 14
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/ml
Arm/Group | Microgynon + Cladribine | Microgynon + Placebo
Number analyzed (Participants) | 21 | 21
pg/ml
  Ethinyl Estradiol | 32.9 (56.9) | 34.1 (52.6)
  Levonorgestrel | 3810 (45.2) | 3830 (46.8)

7. Primary Outcome: Peak-to-Trough Fluctuation Over One Complete Dosing Interval At Steady State (PTF%)
Description: The PTF within complete dosing interval at steady state, calculated as PTF (%) = ([Cmax - Cmin]/Cav) multiplied by 100. Here, Cmin means the minimum plasma concentration, Cmax means the maximum plasma concentration and Cav means the average plasma concentration of drug and metabolite.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post-dose on Day 14
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage fluctuation
Arm/Group | Microgynon + Cladribine | Microgynon + Placebo
Number analyzed (Participants) | 21 | 21
percentage fluctuation
  Ethinyl Estradiol | 220 (28.0) | 213 (23.2)
  Levonorgestrel | 140 (29.7) | 145 (29.0)

8. Secondary Outcome: Number of Participants With Treatment -Emergent Adverse Events (TEAEs)
Description: Adverse event (AE): any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. Serious AE: an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAE: AE with onset after start of treatment or with onset date before the treatment start date but worsening after the treatment start date. TEAEs included both serious and non-serious TEAEs.
Time Frame: Up to Day 84
Population: Safety Analysis Set included all participant who were administered any dose of the trial medication.
Measure: Count of Participants; unit: Participants
Groups:
- Run-in Period: Microgynon (Day -28 to -1): Participants received Microgynon for 21 days, starting on the first day of the menstrual cycle.
- Sequence 1 Period 1: Microgynon Alone (Day 1-8); Sequence 1 Period 2: Microgynon Alone (Day 1-8); Sequence 2 Period 1: Microgynon Alone (Day 1-8); Sequence 2 Period 2: Microgynon Alone (Day 1-8): Participants received a single once daily dose of Microgynon® tablet from Day 1-8.
- Sequence 1 Period 1: Microgynon + Cladribine (Day 9-28): Participants received 5-day once daily dose of Cladribine 10 to 20 milligram(mg) depending on body weight along with Microgynon® tablet once daily from Day 9-28.
- Sequence 1 Period 2: Microgynon + Placebo (Day 9-14): Participants received 5-day once daily dose of Cladribine matched Placebo along with Microgynon® from Day 9-14.
- Sequence 1 Period 2: Microgynon + Cladribine (Day 15-28): Participants received 5-day once-daily dose of Cladribine 10 to 20 mg depending on body weight along with Microgynon® tablet once daily from Day 15-28.
- Sequence 2 Period 1: Microgynon + Placebo (Day 9-28): Participants received 5-day once-daily dose of Cladribine matched Placebo along with Microgynon® from Day 9-28.
- Sequence 2 Period 2: Microgynon + Cladribine (Day 9-28): Participants received 5-day once-daily dose of Cladribine 10 to 20 mg depending on body weight along with Microgynon® tablet once daily from Day 9-28.
Arm/Group | Run-in Period: Microgynon (Day -28 to -1) | Sequence 1 Period 1: Microgynon Alone (Day 1-8) | Sequence 1 Period 1: Microgynon + Cladribine (Day 9-28) | Sequence 1 Period 2: Microgynon Alone (Day 1-8) | Sequence 1 Period 2: Microgynon + Placebo (Day 9-14) | Sequence 1 Period 2: Microgynon + Cladribine (Day 15-28) | Sequence 2 Period 1: Microgynon Alone (Day 1-8) | Sequence 2 Period 1: Microgynon + Placebo (Day 9-28) | Sequence 2 Period 2: Microgynon Alone (Day 1-8) | Sequence 2 Period 2: Microgynon + Cladribine (Day 9-28)
Number analyzed (Participants) | 28 | 13 | 13 | 13 | 13 | 13 | 11 | 10 | 10 | 10
Participants | 7 | 3 | 9 | 5 | 5 | 4 | 1 | 5 | 1 | 7

9. Secondary Outcome: Number of Participants With Clinically Relevant Change From Baseline in Laboratory Values
Description: Laboratory investigation included hematology, biochemistry and urinalysis. Clinical relevance was decided by the investigator. Number of participants with clinically relevant change from baseline in laboratory values were reported.
Time Frame: Up to Day 84
Population: Safety Analysis Set included all participant who were administered any dose of the trial medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Period: Microgynon (Day -28 to -1) | Sequence 1 Period 1: Microgynon Alone (Day 1-8) | Sequence 1 Period 1: Microgynon + Cladribine (Day 9-28) | Sequence 1 Period 2: Microgynon Alone (Day 1-8) | Sequence 1 Period 2: Microgynon + Placebo (Day 9-14) | Sequence 1 Period 2: Microgynon + Cladribine (Day 15-28) | Sequence 2 Period 1: Microgynon Alone (Day 1-8) | Sequence 2 Period 1: Microgynon + Placebo (Day 9-28) | Sequence 2 Period 2: Microgynon Alone (Day 1-8) | Sequence 2 Period 2: Microgynon + Cladribine (Day 9-28)
Number analyzed (Participants) | 28 | 13 | 13 | 13 | 13 | 13 | 11 | 10 | 10 | 10
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Relevant Change From Baseline in Electrocardiogram (ECG)
Description: The 12-lead ECGs were recorded after the participants have rested for at least 5 minutes in supine position. The parameters included heart rate (HR), Respiratory Rate, Pulse Rate, QRS, QT and QTcB calculated by the Bazett formula. Clinical Relevance was decided by the investigator. Number of participants with clinical relevant change from baseline in ECG parameters were reported.
Time Frame: Up to Day 84
Population: Safety Analysis Set included all participant who were administered any dose of the trial medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Period: Microgynon (Day -28 to -1) | Sequence 1 Period 1: Microgynon Alone (Day 1-8) | Sequence 1 Period 1: Microgynon + Cladribine (Day 9-28) | Sequence 1 Period 2: Microgynon Alone (Day 1-8) | Sequence 1 Period 2: Microgynon + Placebo (Day 9-14) | Sequence 1 Period 2: Microgynon + Cladribine (Day 15-28) | Sequence 2 Period 1: Microgynon Alone (Day 1-8) | Sequence 2 Period 1: Microgynon + Placebo (Day 9-28) | Sequence 2 Period 2: Microgynon Alone (Day 1-8) | Sequence 2 Period 2: Microgynon + Cladribine (Day 9-28)
Number analyzed (Participants) | 28 | 13 | 13 | 13 | 13 | 13 | 11 | 10 | 10 | 10
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Relevant Change From Baseline in Vital Signs
Description: Vital signs included oral body temperature, systolic blood pressure, diastolic blood pressure, and pulse rate. Clinical Relevance was decided by the investigator. Number of participants with clinically relevant change from baseline in vital signs were reported.
Time Frame: Up to Day 84
Population: Safety Analysis Set included all participant who were administered any dose of the trial medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Period: Microgynon (Day -28 to -1) | Sequence 1 Period 1: Microgynon Alone (Day 1-8) | Sequence 1 Period 1: Microgynon + Cladribine (Day 9-28) | Sequence 1 Period 2: Microgynon Alone (Day 1-8) | Sequence 1 Period 2: Microgynon + Placebo (Day 9-14) | Sequence 1 Period 2: Microgynon + Cladribine (Day 15-28) | Sequence 2 Period 1: Microgynon Alone (Day 1-8) | Sequence 2 Period 1: Microgynon + Placebo (Day 9-28) | Sequence 2 Period 2: Microgynon Alone (Day 1-8) | Sequence 2 Period 2: Microgynon + Cladribine (Day 9-28)
Number analyzed (Participants) | 28 | 13 | 13 | 13 | 13 | 13 | 11 | 10 | 10 | 10
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Cladribine
Description: Cmax was obtained from plasma concentration time curve.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5 and 2 hours post-dose on Day 10, 11, 12 and 13
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Microgynon + Cladribine
Number analyzed (Participants) | 21
nanogram per milliliter (ng/mL)
  Day 10 | 29.3 (39.4)
  Day 11 | 28.2 (45.5)
  Day 12 | 23.6 (37.5)
  Day 13 | 22.7 (40.7)

13. Secondary Outcome: Time to Reach the Maximum Observed Plasma Concentration (Tmax) of Cladribine
Description: Tmax was obtained from plasma concentration time curve.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5 and 2 hours post-dose on Day 10, 11, 12 and 13
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Microgynon + Cladribine
Number analyzed (Participants) | 21
hours
  Day 10 | 0.500 [0.500 to 1.50]
  Day 11 | 0.500 [0.250 to 1.50]
  Day 12 | 0.500 [0.500 to 1.50]
  Day 13 | 0.500 [0.250 to 2.00]

ADVERSE EVENTS:
Time Frame: Up to Day 84
Arm/Group | Run-in Period: Microgynon (Day -28 to -1) | Sequence 1 Period 1: Microgynon Alone (Day 1-8) | Sequence 1 Period 1: Microgynon + Cladribine (Day 9-28) | Sequence 1 Period 2: Microgynon Alone (Day 1-8) | Sequence 1 Period 2: Microgynon + Placebo (Day 9-14) | Sequence 1 Period 2: Microgynon + Cladribine (Day 15-28) | Sequence 2 Period 1: Microgynon Alone (Day 1-8) | Sequence 2 Period 1: Microgynon + Placebo (Day 9-28) | Sequence 2 Period 2: Microgynon Alone (Day 1-8) | Sequence 2 Period 2: Microgynon + Cladribine (Day 9-28)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/13 | 0/13 | 0/13 | 0/13 | 0/13 | 0/11 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/13 | 0/13 | 0/13 | 0/13 | 0/13 | 0/11 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 7/28 | 3/13 | 9/13 | 5/13 | 5/13 | 4/13 | 1/11 | 5/10 | 1/10 | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Period: Microgynon (Day -28 to -1) (N=28) | Sequence 1 Period 1: Microgynon Alone (Day 1-8) (N=13) | Sequence 1 Period 1: Microgynon + Cladribine (Day 9-28) (N=13) | Sequence 1 Period 2: Microgynon Alone (Day 1-8) (N=13) | Sequence 1 Period 2: Microgynon + Placebo (Day 9-14) (N=13) | Sequence 1 Period 2: Microgynon + Cladribine (Day 15-28) (N=13) | Sequence 2 Period 1: Microgynon Alone (Day 1-8) (N=11) | Sequence 2 Period 1: Microgynon + Placebo (Day 9-28) (N=10) | Sequence 2 Period 2: Microgynon Alone (Day 1-8) (N=10) | Sequence 2 Period 2: Microgynon + Cladribine (Day 9-28) (N=10)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 2 | 0 | 3
Tonsilitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematocrit Decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 6 | 3 | 2 | 3 | 1 | 3 | 0 | 3
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypomenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intermenstrual Bleeding (Reproductive system and breast disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Feeling Cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal Dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Multiple Sclerosis Relapse (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sleep Disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye Pruritus (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation Increased (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood Creatine Phosphokinase MB Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Low Density Lipoprotein Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meralgia Paraesthetica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/44/NCT03745144/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT03745144/SAP_001.pdf